CLINICAL TRIAL: NCT05169372
Title: Retrospective Analysis of 68Ga-PSMA-PET in Patients With Prostate Cancer: Experience From Brazil
Acronym: PET-PSMA
Status: Terminated | Type: Observational
Why Stopped: LACOG and Astellas decided to end the study due to the great difficulty in finding patients with the desired profile.
Sponsor: Latin American Cooperative Oncology Group (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: LACOG 0121
Record Dates: First submitted 2021-12-20; First posted 2021-12-23 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gallium-68-prostate-specific membrane antigen (68Ga-PSMA) positron emission tomography (PET) has been increasingly used in the management of PCa in Brazil. Thus, the detection of metastatic lesions is improved over traditional methods e.g. MRI and the diagnosis of mCSPC patients has been proportionally increasing. Due to a lack of guidelines and clinical trials including 68Ga-PSMA-PET imaging, the management of these patients is extrapolated from data based on conventional imaging. Treatment decision and duration of treatment for mCSPC patients based on 68Ga-PSMA-PET imaging is currently unknown. 68Ga-PSMA-PET allows a diagnosis of a different set of low volume oligo-metastatic prostate cancer patients. Based on that, a new gap has been built up, since there are no standards of how those patients are managed and how they respond to conventional therapies, to metastasis direct therapy or even if they could be spared of any treatment, reducing costs and toxicities. This patient population has not been included in clinical trials and its critical to generate information on the diagnosis, treatment and outcome of these patients in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Age of at least 18 years at study entry;
2. Histologically confirmed adenocarcinoma of the prostate;
3. 68Ga-PSMA-PET exam performed between October 2015 and January 2021;
4. 68Ga-PSMA-PET performed in one of the following situations:

   * localized disease at diagnosis in patients with no detection of extra-prostatic disease in traditional imaging such as CT scan, MRI and bone scan;
   * biochemical recurrence (according to PCWG3 or defined by the investigator) in patients with no detection of prostatic or extra-prostatic disease in traditional imaging such as CT scan, MRI and bone scan;
5. Traditional imaging (pelvic and abdominal CT or MRI and bone scan) with negative results (no extra-prostatic disease, for localized and biochemical recurrence disease; no prostatic for biochemical recurrence disease) performed within 8 weeks before 68Ga-PSMA-PET;
6. Site and investigator ability to collect adequate patient characteristics, treatment and outcome data from medical records.

Exclusion Criteria:

1. Patients with no disease characteristics accessible in medical records;
2. Cancer diagnosis other than prostate cancer in the last 5 years;
3. Disease detected by traditional imaging techniques (bone scan, CT and/or MRI), meaning extra-prostatic disease, for localized and biochemical recurrence disease; or prostatic disease for biochemical recurrence disease.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with localized or biochemical recurrence prostate cancer with no detection of extra-prostatic disease in traditional imaging (bone scan and abdominal and pelvic CT or MRI) who underwent 68Ga-PSMA-PET imaging between October 2015 and January 202.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
The rate of patients with 68Ga-PSMA-PET positive lesions | January 2021
  The rate of patients with 68Ga-PSMA-PET positive lesions [defined as the presence of lesions with 68Ga-PSMA uptake in the prostate (biochemical recurrence) and in extra-prostatic sites (localized disease and biochemical recurrence) in patients with no detected lesions in conventional imaging (no extra prostatic disease, for localized and biochemical recurrence disease; or prostatic disease for biochemical recurrence disease)]

SECONDARY OUTCOMES:
68Ga-PSMA-PET prostate cancer confirmed detection rate | January 2021
  Defined as the proportion of patients with prostate cancer confirmed by histopathology or with PSA response (reduction ≥ 50% on PSA levels from baseline) in those treated with lesion-directed therapy without ADT in day + 90)
Treatment patterns in evaluable patients based on 68Ga-PSMA-PET diagnostic status | January 2021
The percentage of change in initial treatment plan considering the results of 68Ga-PSMA-PET in negative traditional imaging | January 2021
To describe the type of disease monitoring imaging technique (i.e., CT scan, MRI, 68Ga-PSMA-PET) methods after initial diagnosis with 68Ga-PSMA-PET | January 2021
Clinical effectiveness of first-line treatment based on 68Ga-PSMA-PET diagnostic status | January 2021
  (no extra-prostatic disease - localized disease or local recurrence); nodal positive/metastasis negative (regional disease) and metastasis positive (distant disease)
Treatment duration of first-line treatment based on 68Ga-PSMA-PET diagnostic status | January 2021

CONTACTS AND LOCATIONS:
Overall Officials: Andrey Soares, Principal Investigator — Latin American Cooperative Oncology Group
Locations (3):
- Brazil (3):
  - HMV - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - CPO - Centro de Pesquisa em Oncologia do Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Instituto COI - Clínicas Oncológicas Integradas (Instituto Américas RJ), Rio de Janeiro

IPD SHARING:
Plan to Share IPD: No